CLINICAL TRIAL: NCT02784912
Title: Biomarkers-related riSk sTratification of Arrhythmia Recurrence in Patients undergOing Ablation of Sustained ventRicular Tachycardia or Electrical storM - STORM Study
Brief Title: Biomarkers in Risk Stratification of Sustainted Ventricular Tachycardia or Electrical Storm After Ablation
Acronym: STORM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marcin Grabowski, Clinical Professor, Marcin Grabowski, Medical University of Warsaw, Medical University of Warsaw
Other Study IDs: STORM
Record Dates: First submitted 2016-05-21; First posted 2016-05-27 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure; Ventricular Tachycardia; Ventricular Dysfunction
Keywords: Biomarkers; Ventricular Dysfunction; Ventricular Tachycardia; Electrical Storm; ST2; Galectin-3; NT-proBNP; Iron Deficiency; hs-CRP; hs-TnT
MeSH Terms: conditions — Heart Failure; Tachycardia, Ventricular; Ventricular Dysfunction; Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — From each patient will be collected 10 ml of venous blood which will be centrifurgated to obtain serum.
Oversight: Data Monitoring Committee: No

SUMMARY:
Prevalence of HF reaches 1-2% of developed populations, and consequently a significant problem becomes more frequent occurrence of ventricular arrhythmias (VA) - sustained ventricular tachycardia (sVT) and electrical storm (ES) requiring radiofrequency ablation.

The aim of the study is to create a model of risk stratification to identify patients with increased risk of occurrence of composite (cardiovascular death or rehospitalization, arrhythmia recurrence) and secondary (inadequate device therapy, all-cause death or rehospitalization, intensification of atrial arrhythmia) endpoints after ablation of ES or sustained VT. Model will be based on additional measurements of N-terminal pro brain natriuretic peptide (NT-proBNP), Galectin-3, suppressor of tumorigenicity 2 (ST2), high sensitive troponin T (hs-TnT), high sensitive C-reactive protein (hs-CRP), iron deficiency to clinical-, electrocardiographic- and echocardiographic assessment.

DETAILED DESCRIPTION:
Patients with ischemic heart failure (HF) and reduced left ventricle ejection fraction are at high risk for recurrence of VA, ultimately leading to death. Such patients often require ablation. On the other hand, ablation of the VA in patients with post-infarction scar is a technically difficult procedure and often is associated with short-term efficacy.

Risk factors for recurrence of VA are difficult to identify, although there are mentioned e.g. reduced left ventricular ejection fraction, exacerbation of chronic HF and electrolyte abnormalities.

VA is triggered by ongoing inflammation and fibrosis, which are reflected by a level of biomarkers. Thus, it is worth searching for biomarkers that increase the possibility of effective stratification of risk of arrhythmia recurrence in patients undergoing ablation of sVT or ES.

The hypothesis of this study is that biomarker-related risk stratification may be beneficial for patients with ES or sVT.

Sample size assessment was made to specify the number of participants necessary to demonstrate an effect.

The study will include at least 50 patients (who meet the inclusion/exclusion criteria) with ischemic heart failure, with reduced left ventricle ejection fraction admitted to hospital and qualified for ablation due to ES or sVT.

For every patient will be provided case report forms (CRFs) including their clinical status at admission and at discharge, laboratory findings, management during index hospitalization, data from ablation procedure, pharmacotherapy, as well as in-hospital and one-year outcome.

Serum will be collected before ablation and 1-month after discharge from hospital for biomarkers measurements. Patients will be tele-monitored for ≥12-months. There will be carried out two control visits (including assessment of clinical, echocardiographic, electrocardiographic and Holter-ECG parameters) on 1- and 3 months after discharge.

ELIGIBILITY:
Inclusion Criteria (all required):

* >= 18 years
* signed consent
* ischemic heart disease
* left ventricle ejection fraction <= 35%
* admission to hospital due to electrical storm or sustained ventricular tachycardia and qualification for ablation of the arrhythmia
* patients with already implanted cardioverter defibrillator (ICD) / cardiac resynchronization therapy defibrillator (CRT-D) or patients qualified for implantation

Exclusion Criteria:

* non-ischemic heart disease
* current ischemia and potentially reversible causes (e.g. electrolyte abnormalities, drug intoxication) of the arrhythmia
* congenital genetic heart disease
* serious comorbidities (e.g. neoplasm)
* chronic inflammatory disease (e.g. inflammatory bowel disease, rheumatoid arthritis)
* renal failure (creatinine >2,5 mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will include patients with ischemic heart disease with reduced left ventricle ejection fraction admitted to hospital and qualified for ablation due to electrical storm or sustained ventricular tachycardia.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Biomarker-related risk stratification of composite endpoint (cardiovascular death or rehospitalization, arrhythmia recurrence) occurrence after ablation of sustained ventricular tachycardia or electrical storm. | up to 12 months

SECONDARY OUTCOMES:
Biomarker-related risk stratification of secondary endpoint (all-cause death or rehospitalization, intensification of atrial arrhythmia) occurrence after ablation of sustained ventricular tachycardia or electrical storm. | up to 12 months

OTHER OUTCOMES:
Correlation of serum biomarkers concentrations with cardiac remodeling. | up to 12 months
Correlation of serum biomarkers concentrations with hemodynamic stress. | up to 12 months
Assessment of iron deficiency and its prognostic significance. | up to 12 months
Assessment of changes in biomarker levels in serial measurements. | up to 12 months
Correlation of serum biomarkers concentrations in patients with and without device (ICD or CRT-D) already implanted. | up to 12 months
Correlation of serum biomarkers concentrations with a size of an infarct scar. | during index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Marcin D Grabowski, PhD, Study Chair — 1st Department of Cardiology Medical University of Warsaw; Piotr Lodzinski, PhD, Study Chair — 1st Department of Cardiology Medical University of Warsaw; Grzegorz Opolski, Professor, Study Chair — 1st Department of Cardiology Medical University of Warsaw
Locations (1):
- 1st Department of Cariology of Medcial University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
The investigators will be able to share data for meta-analyses